CLINICAL TRIAL: NCT03155867
Title: Plasma Glucose and Insulin Response to Six Meal Replacements in Persons With Type 2 Diabetes Mellitus
Brief Title: Glycemic Response to Six Meal Replacements in Persons With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16.11.US.HCN
Record Dates: First submitted 2017-05-15; First posted 2017-05-16 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-05

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Meal replacement A (Active Comparator)
  Interventions: Other: Meal replacement
- Meal replacement B (Active Comparator)
  Interventions: Other: Meal replacement
- Meal replacement C (Active Comparator)
  Interventions: Other: Meal replacement
- Meal replacement D (Active Comparator)
  Interventions: Other: Meal replacement
- Meal replacement E (Active Comparator)
  Interventions: Other: Meal replacement
- Meal replacement F (Active Comparator)
  Interventions: Other: Meal replacement

INTERVENTIONS:
Other: Meal replacement — The study interventions contain protein, carbohydrate and fat and are intended for use as complete meal replacements for weight loss.

SUMMARY:
This will be a randomized, cross-over design. Subjects will be randomized to one of six interventions on six separate study days, 1 week apart.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-75 yrs
* Type 2 diabetes controlled with diet or diet and oral agent, with the exception of sulfonylureas such as glimepiride (Amaryl), glipizide (Glucotrol/Glucotrol XL) and glyburide (DiaBeta, Micronase, Glynase Prestabs); meglitinides such as reaglinide (Prandin) and nateglinide (Starlix); and alpha-glucosidase inhibitors such as acarbose (Precose) and miglitol (Glyset)
* Hemoglobin A1C less than 9.0%
* Fasting blood glucose less than 180 mg
* Hematocrit levels within normal limits

Exclusion Criteria:

* Abnormal thyroid function
* Creatinine >2.0 mg/dL
* Potassium <3.5 mEq/L
* Gastrointestinal disease: ulcer, gastritis, diarrhea, gastroparesis, vomiting
* Currently unstable diabetes or under treatment for cancer, heart disease, renal disease
* Unable to give informed consent or follow instructions
* Current insulin therapy or insulin therapy within the past month
* Patient who are pregnant
* Allergies to milk, soy or any component of the test product
* Patient who in the Investigators assessment cannot be expected to comply with treatment
* Currently participating or having participated in another clinical trial.
* Patients with Anemia

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2017-05-18 (Actual); Study Completion 2017-05-18 (Actual)

PRIMARY OUTCOMES:
Area under the blood glucose curve (AUC 0-240) | Baseline, 10, 20, 30, 60, 90, 120, 150, 180, 210 and 240 minutes

SECONDARY OUTCOMES:
Area under the insulin curves (AUC 0-240) | Baseline, 10, 20, 30, 60, 90, 120, 150, 180, 210 and 240 minutes
Insulinogenic index [Change in Ins30/Change in Glu30] | Baseline, 10, 20, 30, 60, 90, 120, 150, 180, 210 and 240 minutes
AUC (0-30min) for insulin | Baseline, 10, 20, 30, 60, 90, 120, 150, 180, 210 and 240 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Joel Neutel, MD, Principal Investigator — Orange County Research Center
Locations (1):
- Orange County Research Center, Tustin, California, United States